CLINICAL TRIAL: NCT04938466
Title: Assessment of Adherence, Quality of Life, Clinical Response and Safety of Daily and Long-Acting Growth Hormone Therapy
Acronym: LAuGH TRACK
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2020-28945
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Growth Hormone Deficiency; Growth Hormone Treatment
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum samples for Growth Hormone Antibodies will be stored in the freezer storage of the M Health Fairview University of Minnesota Medical Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Transition to long-acting growth hormone (LAGH): Participants in this arm will transition between daily growth hormone treatment and long-acting growth hormone treatment.
  Interventions: Drug: Long-Acting Growth Hormone (LAGH)
- Consistent daily growth hormone (DGH): Participants in this group will continue with daily growth hormone treatment.

INTERVENTIONS:
Drug: Long-Acting Growth Hormone (LAGH) — Long-acting growth hormone (LAGH) treatment
  Groups: Transition to long-acting growth hormone (LAGH)

SUMMARY:
The purpose of the study is to compare quality of life, adherence, insulin resistance, body composition and efficacy of long-acting growth hormone (LAGH) to daily growth hormone (DGH) in children with growth hormone deficiency (GHD). These objectives will be evaluated every 6 months for subjects prior to switch from DGH to LAGH, and 6 months after.

DETAILED DESCRIPTION:
Daily subcutaneous injections of recombinant human growth hormone (GH) is the standard of care therapy for children with GH deficiency (GHD). A potential impediment to long-term efficacy of daily GH (DGH) is a lack of adherence and persistence. Multiple Long-Acting Growth Hormone (LAGH) molecules are being developed with the expectation that reduced frequency of injections will improve the patient and caregiver experience leading to improved adherence and, ultimately, improve efficacy. However, the connection between reduced injection frequency, improved adherence and improved efficacy have not yet been demonstrated. GH has metabolic effects that impact insulin resistance, body composition and lipid levels. There is concern that persistently elevated levels of GH provided by LAGH may have a negative effect on metabolism. There is also concern that the larger size of the LAGH molecules in development may limit their access to the target tissues leading to an imbalance of the linear growth and metabolic effects. The purpose of the study is to compare quality of life, adherence, insulin resistance, body composition and efficacy of long-acting growth hormone (LAGH) to daily growth hormone (DGH) in children with growth hormone deficiency (GHD). These objectives will be evaluated every 6 months for subjects prior to switch from DGH to LAGH, and 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* Girls must be between the ages of 2 and 11 years, and boys must be between the ages of 2 and 13 years
* Have established diagnosis of pediatric growth hormone deficiency (GHD). For the purposes of the study, GHD is defined as peak growth hormone response to clonidine/arginine stimulation testing of <10 ng/mL
* Either treatment-naive or currently treated with a daily growth hormone as approved by health insurance

Exclusion Criteria:

* Any medical condition which, in the opinion of the Investigator, can be an independent cause of short stature and/or limit the response to exogenous growth factor treatment
* Current treatment with long-acting growth hormone
* Currently pregnant or breastfeeding

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving daily growth hormone treatment for growth hormone deficiency (GHD).
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Resistance | Every six months for approximately 2 years
  Fasting glucose and insulin will be measured using standard laboratory tests in order to calculate homeostatic model assessment of insulin resistance (HOMA-IR). The equation is as follows, fasting plasma glucose (mmol/l) multiplied by fasting serum insulin (mU/l) divided by 22.5. HOMA-IR is a unitless measure with no defined range. Higher scores indicate lower insulin sensitivity/higher insulin resistance. Insulin resistance will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Bone Mineral Density - DXA | Every six months for approximately 2 years
  Bone mineral density will be measured using dual energy X-ray absorptiometry (DXA) reported in units of grams per centimeter^2. Bone density will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Bone Mineral Density - pQCT | Every six months for approximately 2 years
  Bone mineral density will be measured using peripheral quantitative computed tomography (pQCT) and reported in units of grams per centimeter^3. Bone density will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Percent Fat | Every six months for approximately 2 years
  Percent fat will be measured using dual energy X-ray absorptiometry (DXA), peripheral quantitative computed tomography (pQCT), and BodPod and reported in units of percent kilograms. Percent fat will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Fat Free Mass | Every six months for approximately 2 years
  Fat free mass will be measured using dual energy X-ray absorptiometry (DXA), peripheral quantitative computed tomography (pQCT), and BodPod and reported in units of kilograms. Fat free mass will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Muscle Content - DXA | Every six months for approximately 2 years
  Muscle content will be measured using dual energy X-ray absorptiometry (DXA) and BodPod and reported in units of percent kilograms. Muscle content will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in Muscle Content - pQCT | Every six months for approximately 2 years
  Muscle content will be measured using peripheral quantitative computed tomography (pQCT) and reported in units of grams per centimeter^3. Muscle content will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.

SECONDARY OUTCOMES:
Change in PedsQL Questionnaire | Every six months for approximately 2 years
  The PedsQL Questionnaire contains 23 items rated on a 3- or 5-point Likert scale. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Total score is calculated as the unweighted average of item scores. Higher scores indicate better health-related quality of life. PedsQL will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in QOLISSY Questionnaire | Every six months for approximately 2 years
  The QOLISSY Questionnaire contains 66 items rated on a 5-point Likert scale. Total score is calculated as the mean of item scores. Total scores range from 66 to 330 with higher scores indicating better quality of life. QOLISSY will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in DID-EQ Questionnaire | Every six months for approximately 2 years
  The Diabetes Injection Device - Experience Questionnaire (DID-EQ) contains 10 items on a 4-point Likert scale. Total score is calculated as a weighted average of item scores. Total scores range from 10 to 40 with higher score indicating more positive perceptions of injection device characteristics. DID-EQ will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.
Change in DID-PQ Questionnaire | Every six months for approximately 2 years
  The Diabetes Injection Device - Preference Questionnaire (DID-EQ) contains 10 items on a 5-point Likert scale (-2 to 2), with a total range of -20 to 20. Scores on each end of the scale equal a more positive perception of the device. A higher score indicates a stronger preference for LAGH device and a lower (negative) score indicates a preference for daily growth hormone device. Results will be reported descriptively and categorically as the frequency and percentage of patients reporting each response to each item. DID-EQ will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to
Change in Adherence Survey | Every six months for approximately 2 years
  An adherence survey will be administered and medication possession ratio (MPR) data will be obtained. Likert scale items will be measured with a range of 26 to 121, with a higher score indicating a greater burden to growth hormone treatment. Non-Likert scale items (2 items with percent report and 2 items with Yes/No responses) will not be added to a total score but will be reported descriptively. Adherence will be assessed at baseline, 6 months prior to beginning LAGH treatment, and 6 months following the start of LAGH treatment, or every 6 months for two years for those who do not switch to LAGH. Change in values will be reported, for participants on Daily Growth Hormone who never switch to LAGH, from baseline to values obtained at 6 months, 12 months, 18 months, and 24 months. For participants who switch to LAGH, baseline values pre-LAGH treatment will be compared to those obtained 6 months following the start of LAGH treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Miller, MD, PhD, Principal Investigator — University of Minnesota Department of Pediatric Endocrinology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No